CLINICAL TRIAL: NCT01265810
Title: Phase III Randomized Double-blind Cross-over Trial of Caphosol® Versus NaCl 0.9% in the Relief of Oral Mucositis in Renal Cell Carcinoma, Hepatocellular Carcinoma, and Gastrointestinal Stromal Tumor Patients Receiving Targeted Therapy
Brief Title: Caphosol in Oral Mucositis Due to Targeted Therapy
Acronym: COMTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impaqtt Foundation (Other)
Collaborators: CB Boers ORG (Other); Memorial Sloan Kettering Cancer Center (Other); Leiden University Medical Center (Other); Pfizer (Industry); Novartis (Industry); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Impaqtt-002
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Oral Complaints; Renal Cell Carcinoma; Hepatocellular Carcinoma; Gastrointestinal Stromal Tumors
Keywords: stomatitis; targeted therapy; Caphosol; mouthrinses
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Gastrointestinal Stromal Tumors; Stomatitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sodium chloride -> supersaturated calcium-phosphate (Other): Patients in this arm start first with sodium chloride 0.9% mouth rinses and go crossover to supersaturated calcium-phosphate mouth rinses.
  Interventions: Other: supersaturated calcium-phosphate; Other: sodium chloride 0.9 %
- supersaturated calcium-phosphate -> sodium chloride (Other): Patients in this arm start first with supersaturated calcium-phosphate mouth rinses and go crossover to sodium chloride 0.9% mouth rinses.
  Interventions: Other: supersaturated calcium-phosphate; Other: sodium chloride 0.9 %

INTERVENTIONS:
Other: supersaturated calcium-phosphate — 4 times daily, 2 minutes rinse with 30 ml solution during active rinse period (14 days)
  Other Names: Caphosol
Other: sodium chloride 0.9 % — 4 times daily, 2 minutes rinse with 30 ml solution during active rinse period (14 days)

SUMMARY:
Targeted therapies such as multi-targeted tyrosine kinase inhibitors (TKI) and mammalian target of rapamycin inhibitors (mTORI) in renal cell carcinoma (RCC), demonstrate a high level of efficacy with acceptable tolerability. Currently, there are five approved targeted therapies available for RCC: sunitinib (Sutent®), sorafenib (Nexavar®), pazopanib (Votrient®), temsirolimus (Torisel®), and everolimus (Afinitor®). Hepatocellular carcinoma treated with sorafenib and gastro intestinal stromal tumors patients treated with sunitinib will be included, too.

Since this agents have dermatological adverse events in common, with oral mucositis (OM), hand-foot skin reaction (HFSR) and papulopustular eruption (PPE) as an disabling side effect, we require evidence based management options to prevent and treat these adverse events. The incidence of OM of any grade is for sunitinib 38%, sorafenib 28%, pazopanib 4%, temsirolimus 41%, and everolimus 44%. Recent data suggest that TKI and mTORI associated OM is distinct from conventional mucositis and more closely resembles aphthous OM.

Recently, supersaturated calcium-phosphate rinse (Caphosol®), a Ca2+/PO43- mouth rinse, became available to prevent or treat OM.

The objective is to assess the relieving effect of Caphosol® oral rinse on clinical outcomes which include oral intake, swallowing function and pain associated with incidence of grade ≥ 1 oral side effects and the anticancer therapy cessation in patients treated with selected targeted anticancer therapy.

Patients with OM > grade 0 on targeted therapy will be randomly allocated to receive either Caphosol® or NaCl 0.9% rinse for two weeks. After the first rinse period all patients will switch to the opposite treatment arm (NaCl 0.9% or Caphosol®) for another two weeks. Duration of oral side effects, severity, pain, dose of analgesics and tolerability will be assessed weekly with the Modified-VHNSS-version-2.0 oral-specific questionnaire. Patients will be stratified by targeted anticancer agent and per tumor type (pre-defined cohorts). Objective severity of oral side effects will be assessed using the NCI-CTCAE v4.0. Correlation of subjective Modified-VHNSS-version-2.0 scores with the objective NCI-CTCAE grade, sex, age, targeted therapy type, and cancer type will be conducted.

DETAILED DESCRIPTION:
OM with mucosal change, associated pain, and taste change - are clinically relevant toxicities of TKI's and mTORI's presently in use. The incidence of oral mucositis of any grade is for sunitinib 38%, sorafenib 28%, pazopanib 4%, temsirolimus 41%, and for everolimus 44%.

Optimal antitumor activity requires maintaining the highest tolerable dose in individual patients. In order to improve health related quality of life (HRQoL) and patient adherence, adverse effects should be prevented, if possible avoided and treated if necessary. Current oral formulations consist of various schedules (continuous administration or 4 weeks on, 2 weeks off) to optimize the benefit-risk profile. Adherence to anti-cancer treatment is particularly important when prescribing oral therapies as adherence to the protocol can have a significant impact on efficacy and the severity of treatment-related AEs. As sorafenib, sunitinib, pazopanib, and everolimus are taken in the outpatient setting, patient education on the correct treatment dosing, usage and the nature, recognition, and severity of AEs is essential.

Recent data suggest that TKI and mTORI associated OM is different from conventional chemotherapy related OM. Oral ulceration usually presents as aphthous-like ulcerations and has in some studies been reported as mucositis. An analysis of the appearance, course, and toxicity experiences demonstrated that the condition is distinct from conventional mucositis and more closely resembles aphthous oral mucositis. These TKI/mTORI related ulcers may represent a dose-limiting toxicity for this new class of agents, especially considering the fact that even lower grade mucositis with chronic daily dosing may be cumbersome to the patient and lead to dose reductions. Studies of treatment strategies for aphthous OM may therefore be important for the dose adherence of TKI and mTORI and for the overall acceptance of this therapy for patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* ≥18 years of age
* Histological proof of RCC, HCC or GIST
* Oral adverse events > grade 0 due to sunitinib, sorafenib, pazopanib, temsirolimus, or everolimus in mono therapy at study entry
* Written informed consent
* Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2
* Able to perform oral rinsing
* Able to complete questionnaires by themselves or with assistance

Exclusion Criteria:

* Any previous systemic antineoplastic treatment within 4 weeks of initiation of current targeted anticancer therapy
* Current antineoplastic combination cytotoxic chemotherapy therapy
* Physiologic condition that precludes the use of an oral rinse
* Hypersensitivity to Caphosol ingredients
* Use of palifermin, oral cryotherapy, low level laser therapy, topical oral steroids within 3 weeks of current targeted anticancer therapy
* Oral abnormalities defined as baseline oral assessment of NCI-CTCAE v4.0 grade > 0
* Current use of agents that are known to be strong inducers or inhibitors of CYP3A4 that can not be stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Assess the severity of patient-reported oral adverse events as determined by the change in the Modified-VHNSS2.0 score 3 times a week, from onset of oral adverse events during the active oral rinse period with Caphosol versus NaCl 0.9% | 2 times 14 days

SECONDARY OUTCOMES:
Determine the decrease in grade of oral adverse events as measured by the NCI-CTCAE v4.0 once a week, during a 2 week treatment with Caphosol oral rinse versus NaCl 0.9% oral rinse, 4 times daily, 2 minutes with 30 ml solution | 2 times 14 days
Assess the incidence of dose delay or dose interruption, dose reduction and discontinue treatment owing to oral burden due to targeted anticancer therapy during the active oral rinse period, once a week | 2 times 14 days
To correlate the incidence of oral mucositis with: grade ≥ 2 hand-foot skin reaction (HFSR), and grade ≥ 2 papulopustular eruption (PPE) with all agents as measured by the NCI-CTCAE v4.0, during the active oral rinse period, once a week | 2 times 14 days
Side Study: Explorative analysis of polymorphism in genes encoding for pharmacokinetic and pharmacodynamic variables related to the pharmacodynamics of the TKIs | once

CONTACTS AND LOCATIONS:
Overall Officials: Christine B. Boers-Doets, MSc, Principal Investigator — CB Boers ORG; Mario E Lacouture, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Hans Gelderblom, MD, PhD, Study Chair — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - The Netherlands Cancer Institute-Antoni van Leeuwenhoek Hospital, Amsterdam
  - Leiden University Medical Centre (LUMC), Leiden